CLINICAL TRIAL: NCT02790372
Title: The Effect of Comprehensive Geriatric Assessment and Case Conferencing on Neuropsychiatric Symptoms Among Patients in Norwegian Nursing Homes
Brief Title: The Effect of Case Conferencing in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/1642
Record Dates: First submitted 2016-05-31; First posted 2016-06-03 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2017-04

CONDITIONS: Dementia; Neurobehavioral Manifestations
Keywords: Nursing homes; Norway
MeSH Terms: conditions — Dementia; Neurobehavioral Manifestations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control nursing homes (No Intervention): Nursing homes carries out usual care
- Intervention nursing homes (Active Comparator): Nursing homes that carries out regularly case conferencing
  Interventions: Other: Case conferencing

INTERVENTIONS:
Other: Case conferencing — Intervention nursing homes carries out regularly case conferencing based on comprehensive geriatric assessments. Case conferencing is carried out each month for nursing home patients included in the study
  Arms: Intervention nursing homes

SUMMARY:
This study evaluates the effect of using comprehensive geriatric assessment in combination with case conferences on the prevalence of neuropsychiatric symptoms (also known as behavioral and psychological symptoms of dementia) in Norwegian nursing homes

DETAILED DESCRIPTION:
Long-term care patients in nursing homes (NH) are characterized by frailty and having multiple health problems and reduced quality of life. Some of these issues relates to the quality of care and do therefore possess a potential for improvement. There is a need for approaches enabling nurses to carry out effective interventions that can promote health related to sustain or improve the nursing home patients health status. Integrating a comprehensive geriatric assessment (CGA) and case conferencing (CC) might be an effective method to individualize care plans in order to improve quality of care.

The intervention nursing homes will implement CGA, using the International resident instrument suite for Long Term Care Facilities (InterRai LTCF) and CC. The patients will be included and assessed three times during a 12-month period (control and intervention NHs). In the intervention NHs the results from the CGA will be reviewed in monthly CCs. The CCs are structured and consist of four main steps; evaluating the effects of earlier interventions, defining patients risks or area for improvement, defining the aetiology of the risk or problem, defining interventions and measures for improvement along with an appropriate method for evaluation. The CC group's consensus is basis for the patient's care plan.

ELIGIBILITY:
Inclusion Criteria:

* registered as long term care patient
* been in the nursing home for more than a month
* Informed consent from the patient or legal guardians

Exclusion Criteria:

* life expectancy less than six months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 309 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of neuropsychiatric symptoms measured by neuropsychiatric inventory | 12 months
  Measured by neuropsychiatric inventory

SECONDARY OUTCOMES:
Depression measured by Cornell scale for depression in dementia | 12 months
  Measured by Cornell scale for depression in dementia
Activities in daily living measured by Physical self-maintenance scale | 12 months
  Measured by Physical self-maintenance scale
Quality of life measured by the Quality of Life in Late-Stage Dementia Scale | 12 months
  Measured by the Quality of Life in Late-Stage Dementia Scale

CONTACTS AND LOCATIONS:
Overall Officials: Sigrid Nakrem, phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Overhalla sykeheim, Overhalla, Norway

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Nakrem S, Stensvik GT, Skjong RJ, Ostaszkiewicz J. Staff experiences with implementing a case conferencing care model in nursing homes: a focus group study. BMC Health Serv Res. 2019 Mar 27;19(1):191. doi: 10.1186/s12913-019-4034-0. PMID 30917815
- [Derived] Stensvik GT, Helvik AS, Haugan G, Steinsbekk A, Salvesen O, Nakrem S. The short-term effect of a modified comprehensive geriatric assessment and regularly case conferencing on neuropsychiatric symptoms in nursing homes: a cluster randomized trial. BMC Geriatr. 2022 Apr 11;22(1):316. doi: 10.1186/s12877-022-02976-x. PMID 35410145